CLINICAL TRIAL: NCT05079243
Title: Examining the Best Solution for Dermal and Subcutaneous Augmentation and Regeneration Using Ex-vivo Expanded Autologous Adipose-derived Stromal Cells, Autologous Fat Tissue and Natural Tissue Scaffolds
Brief Title: Dermal and Subcutaneous Augmentation and Skin Assessment After Fat-, Stem Cell and Scaffold Injections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stemform (Industry)
Collaborators: Rigshospitalet, Denmark (Other); Aleris-Hamlet Hospitaler København (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: H-21004160
Record Dates: First submitted 2021-06-06; First posted 2021-10-15 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Augmentation; Reconstruction

STUDY DESIGN:
Intervention Model Description: Triple blinded, randomized, paired study on healthy participants
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scaffold and adipose-derived stromal cell enriched fat grafts (Experimental): Randomized and paired injections. Each participant will receive all 11 solutions.
  Interventions: Biological: Scaffold and adipose-derived stromal cell enriched fat grafts
- Controls samples (No Intervention): Control samples of untreated skin

INTERVENTIONS:
Biological: Scaffold and adipose-derived stromal cell enriched fat grafts — eight different solutions of fat, ASCs, scaffold and CO2 laser in dermis three different solutions of fat, ASCs and scaffold in the subcutaneous layer
  Arms: Scaffold and adipose-derived stromal cell enriched fat grafts

SUMMARY:
Investigate the effect of dermal/subcutaneous injection of ASC enriched fat transplant in a protective natural scaffold, designed to sustain the ASC viability after dermal/subcutaneous injection.

DETAILED DESCRIPTION:
The study investigates the effect of different concentrations of autologous ex-vivo expanded adipose-derived stromal cells (ASCs), fat and a natural scaffold for skin rejuvenation and augmentation. The aim is to better the volume of fat grafts for cosmetic and reconstructive purposes. Fat is a near ideal filler, as it is biocompatible. However the retention rate of fat grafts often result in poor outcomes and it is unpredictable. The investigators have set up an experimental study in which participants with excess abdominal skin is recruited. They will have injections with 11 different solutions of fat, ACSs, scaffold and dermal CO2 laser in the abdominal skin. After 3 months biopsies will be taken and after 6 months all of the treated area will be removed by an cosmetic abdominoplasty.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18-30 kg/m2
* 400 mL of fat (lipoaspirate) available for liposuction in the thighs or back
* Desire for abdominoplasty
* Speaks and reads Danish
* Signed informed consent

Exclusion Criteria:

* Smoking
* Previous major abdominal surgery
* Previous cancer or predisposition to cancer
* Pregnancy or planned pregnancy
* Known chronic disease associated with metabolic malfunction or poor healing
* Pacemaker
* Allergy to necessary anaesthesia
* Intention of significant weight loss or weight gain within the trial period

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Volume assessment | Baseline, three months, Six months
  CT scan

SECONDARY OUTCOMES:
Cell count, immunohistochemistry, skin quality | Three months, six months
  Cell count, immunohistochemistry, skin quality
Immunohistochemistry | Three months, six months
  Immunohistochemistry
Skin thickness | Three months, six months
  Skin thickness

CONTACTS AND LOCATIONS:
Overall Officials: Frederik P Mamsen, Principal Investigator — StemMedical A/S; stig-Frederik T Koelle, MD, PhD, Principal Investigator — StemMedical A/S
Locations (2):
- Denmark (2):
  - Aleris Hamlet, Copenhagen, Søborg
  - StemMedical, Copenhagen, Søborg

IPD SHARING:
Plan to Share IPD: No
Upon request IPD can be shared with different parties if assessed valid by the primary investigators